CLINICAL TRIAL: NCT01690988
Title: The Prevention of Delirium and Complications Associated With Surgical Treatments Multi Center Clinical Trial
Acronym: PODCAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Asan Medical Center (Other); Weill Medical College of Cornell University (Other); Harvard Medical School (HMS and HSDM) (Other); Medical College of Wisconsin (Other); Memorial Sloan Kettering Cancer Center (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); University of Bern (Other); University of Michigan (Other); University of Manitoba (Other); University Health Network, Toronto (Other); Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Principal Investigator, Michael Avidan, Director, Institute of Quality Improvement, Research & Informatics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201206071
Record Dates: First submitted 2012-08-07; First posted 2012-09-24 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-11

CONDITIONS: Delirium
Keywords: Delirium; ketamine; surgery; neurological complications
MeSH Terms: conditions — Delirium | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketamine (0.5 mg/kg) (Experimental): Low dose (sub-anesthetic) 0.5 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Interventions: Drug: Ketamine (0.5 mg/kg)
- Normal saline (placebo) (Placebo Comparator): Intravenous normal saline
  Interventions: Drug: Normal Saline (placebo)
- Ketamine (1 mg/kg) (Experimental): Low dose (sub-anesthetic) 1 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Interventions: Drug: Ketamine (1 mg/kg)

INTERVENTIONS:
Drug: Ketamine (0.5 mg/kg) — Low dose (sub-anesthetic) 0.5 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Other Names: Ketalar
  Arms: Ketamine (0.5 mg/kg)
Drug: Normal Saline (placebo) — Normal saline IV following induction of anesthesia or administration of sedative medications
  Other Names: Normal saline
  Arms: Normal saline (placebo)
Drug: Ketamine (1 mg/kg) — Low dose (sub-anesthetic) 1 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Other Names: Ketalar
  Arms: Ketamine (1 mg/kg)

SUMMARY:
Delirium is a medical term or condition that includes a temporary inability to focus attention and to think clearly. Delirium occurs commonly (10% to 70%) in patients older than 60 undergoing large surgeries. The purpose of this study is to test rigorously whether a drug called ketamine can decrease the chance that patients will experience delirium after their surgery. The investigators are also testing whether ketamine decreases postoperative pain, postoperative opioid consumption, postoperative nausea and vomiting, ICU and hospital length of stay, and adverse outcomes (e.g. hallucinations and nightmares).

DETAILED DESCRIPTION:
Postoperative delirium is one of the most common complications of major surgery, affecting between 10% and 70% of all elderly surgical patients. Delirium manifests as poor attention and inability to think logically, and is associated with longer intensive care unit and hospital stay, long lasting cognitive deterioration, and increased mortality rate. Studies have shown that a low sub-anesthetic dose of ketamine, an anesthetic drug, has the potential to decrease several postoperative complications, including delirium, pain, opioid consumption, and nausea and vomiting. Low dose ketamine would be particularly appealing as a drug to prevent delirium and other postoperative complications, as it is inexpensive and extremely safe. However, these proposed benefits of ketamine in the perioperative setting have not yet been tested in a large clinical trial. The investigators are therefore proposing a pragmatic, exploratory clinical trial to support or refute the contention that low dose ketamine decreases the incidence of postoperative delirium, with the possibility of conducting a larger randomized clinical trial pending the results of this study. At the time of enrollment, patients will undergo the same delirium and pain evaluation that will be used postoperatively. Additionally patients will be screened for functional dependence using the Barthel Index of Activities of Daily Living, for depression using the Geriatric Depression Scale - Short Form, and for obstructive sleep apnea using the STOP-Bang criteria. They will also be asked about any falls they have experienced in the six months prior to surgery. Comorbid conditions, including the components of the Charlson Comorbidity Index, will be obtained by reviewing the patients' medical records. Any available preoperative lab results, including electrolytes and blood counts, will also be recorded.

Patients will be randomized to receive low dose ketamine or placebo following induction of anesthesia and prior to surgical incision. Blinded observers will assess delirium on the afternoon/evening of postoperative day 0 (if feasible) and twice daily (morning and afternoon/evening with at least six hours between assessments) on postoperative days 1-3 using the Confusion Assessment Method or the Confusion Assessment Method for Intensive Care Unit. Acute pain will be assessed via the observer-based Behavioral Pain Scale or Behavioral Pain Scale (Non-Intubated) with subsequent administration of the patient-reported Visual Analog Scale from postoperative days 0-3. Postoperative opioid consumption will be assessed from the patients' medical charts for postoperative days 0-3. Postoperative nausea and vomiting will be assessed via a patient-reported section of the Behavioral Pain Scale or Behavioral Pain Scale (Non-Intubated) for postoperative days 0-3. ICU and/or hospital length of stay will be assessed from the patients' medical charts. Adverse outcomes (e.g. hallucinations and nightmares) will be assessed via the Confusion Assessment Method or the Confusion Assessment Method for Intensive Care Unit for postoperative days 0-3.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 and older
* Competent to provide informed consent
* Undergoing major surgery (e.g., open cardiac surgery, open or thoracoscopic thoracic surgery, abdominal surgery, open urological surgery, open gynecological surgery, major orthopedic surgery, major vascular surgery including endovascular procedures, major ear, nose and throat surgery).

Exclusion Criteria:

* Patients with an allergy to ketamine
* Those in whom a significant elevation of blood pressure would constitute a serious hazard (e.g., pheochromocytoma, aortic dissection)
* Unable to provide informed consent
* Patients with drug misuse history (e.g., ketamine, cocaine, heroin, amphetamine, methamphetamine, MDMA, phencyclidine, lysergic acid, mescaline, psilocybin)
* Patients taking anti-psychotic medications (e.g., chlorpromazine, clozapine, olanzapine, risperidone, haloperidol, quetiapine, risperidone, paliperidone, amisulpride, sertindole)
* Patients with a weight outside the range 50 kg - 200 kg (110 lbs - 440 lbs)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-06-26 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Mashour, MD PhD, Principal Investigator — University of Michigan; Daniel A Emmert, MD PhD, Study Director — Washington University School of Medicine; Kane Pryor, MBBS, Study Director — Cornell; Eric Jacobsohn, MB ChB, Study Director — University of Manitoba; Judith Hudetz, PhD, Study Director — Medical College of Wisconsin; Hilary P Grocott, MD, Study Chair — University of Manitoba; Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine; Sharon Inouye, Study Director — Harvard Medical School (HMS and HSDM); Robert Veselis, Study Director — Memorial Sloan Kettering Medical Center; Jayant Aveek, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh; Heiko Kaiser, Study Director — University of Bern; Stephen Choi, Study Chair — University of Toronto; Ryan Pong, Study Chair — Virginia Mason Medical Center; Gyujeong Noh, Study Director — Asan Medical Center
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Avidan MS, Fritz BA, Maybrier HR, Muench MR, Escallier KE, Chen Y, Ben Abdallah A, Veselis RA, Hudetz JA, Pagel PS, Noh G, Pryor K, Kaiser H, Arya VK, Pong R, Jacobsohn E, Grocott HP, Choi S, Downey RJ, Inouye SK, Mashour GA. The Prevention of Delirium and Complications Associated with Surgical Treatments (PODCAST) study: protocol for an international multicentre randomised controlled trial. BMJ Open. 2014 Sep 17;4(9):e005651. doi: 10.1136/bmjopen-2014-005651. PMID 25231491
- [Result] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Derived] Vlisides PE, Thompson A, Kunkler BS, Maybrier HR, Avidan MS, Mashour GA; PODCAST Research Group. Perioperative Epidural Use and Risk of Delirium in Surgical Patients: A Secondary Analysis of the PODCAST Trial. Anesth Analg. 2019 May;128(5):944-952. doi: 10.1213/ANE.0000000000004038. PMID 30768457
- [Derived] Mashour GA, Ben Abdallah A, Pryor KO, El-Gabalawy R, Vlisides PE, Jacobsohn E, Lenze E, Maybrier HR, Veselis RA, Avidan MS; PODCAST Research Group. Intraoperative ketamine for prevention of depressive symptoms after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Br J Anaesth. 2018 Nov;121(5):1075-1083. doi: 10.1016/j.bja.2018.03.030. Epub 2018 Sep 19. PMID 30336852

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 746 participants were consented to the study; however only 672 were randomly assigned as 74 participants were determined ineligible after consent. Reasons for ineligibility: operations were cancelled or patients withdrew from the study, etc.
Groups:
- Ketamine (1 mg/kg): High dose (sub-anesthetic) 1 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Ketamine (1 mg/kg): High dose (sub-anesthetic) 1 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
Period: Overall Study
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Started | 227 | 222 | 223
Completed | 221 | 217 | 216
Not Completed | 6 | 5 | 7
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Operation Cancelled | 1 | 1 | 0
Not completed — Determined ineligible | 1 | 0 | 0
Not completed — Death | 1 | 1 | 1
Not completed — Sedated | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg) | Total
Number analyzed (Participants) | 227 | 222 | 223 | 672
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 59 | 61 | 176
  >=65 years | 171 | 163 | 162 | 496
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70 (7.2) | 70 (6.9) | 70 (7.3) | 70 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 87 | 84 | 254
  Male | 144 | 135 | 139 | 418
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 147 | 147 | 149 | 443
  Canada | 63 | 61 | 59 | 183
  India | 6 | 5 | 5 | 16
  South Korea | 11 | 9 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Incidence of Delirium Across All Patients at Baseline and Over Post-operative Days 1-3
Description: According to Confusion Assessment Method or Confusion Assessment Method for Intensive Care Unit criteria the number of patients that had any positive CAM on any day for all patients. The main effect evaluated will be to determine whether ketamine decreases delirium, table 3 of the protocol provides a useful guide for the potential findings of the current study with their implications.
  To further clarify, delirium will be assessed on the day of surgery, when possible and on the subsequent three days POD 1-3, as long as as patients remain in the hospital and are assessable (i.e., not sedated to a RASS <-3). The assessments on POD 1-3 will be done twice daily, once in the morning and once in the afternoon. The primary outcome of the study includes only the delirium incidence on POD 1-3.
  The primary comparison will be between the combined ketamine groups and the placebo group.
Time Frame: Delirium incidence on postoperative days 1-3, calculated by any positive CAM on any day for all patients
Population: Of all 672 participants, data were analyzed AM and PM and post operative day 1 through day 3 for screened participants with a CAM. The overall incidence of delirium were compared, Ketamine 0.5 mg/kg and 1 mg/kg groups were combined as per-specified in the study protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Ketamine (0.5 mg/kg and 1 mg/kg): Both the 0.5 mg/kg and the 1mg/kg doses groups of Ketamine were combined for analysis)
  Low dose Ketamine (sub-anesthetic) 0.5 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Ketamine (1 mg/kg): (sub-anesthetic) 1 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
Arm/Group | Ketamine (0.5 mg/kg and 1 mg/kg) | Normal Saline (Placebo)
Number analyzed (Participants) | 438 | 217
Participants | 85 | 43
Statistical Analysis 1: Comparison: Ketamine (0.5 mg/kg and 1 mg/kg) vs Normal Saline (Placebo); The primary analysis was a comparison between the placebo control group and the combined ketamine groups; Test type: Other — Test of independence; p = 0.912, Chi-squared; Difference in Percentages = 0.36, 95% CI 2-sided [-6.07 to 7.38], Standard Error of Mean 3.301 — Difference in delirium incidence between placebo control and combined ketamine groups

2. Secondary Outcome: Daily Maximum Pain Recorded
Description: Assessed by observer-based Behavioral Pain Scale or Behavioral Pain Scale (Non-Intubated) with subsequent administration of patient-reported Visual Analog Scale The behavioral pain scale has three domains and ranges from 3 to 15. The visual analog scale is a continuous scale from 0 to 100 mm. Daily Maximum Pain accounted for pain level in the AM or PM for both the VAS and the BPS/BPS-NI a higher value means a worse outcome.
Time Frame: Postoperative days 1-3, two assessment daily (morning and afternoon), with at least six hours between assessments
Measure: Median (Inter-Quartile Range); unit: participants
Groups:
- Ketamine (0.5 mg/kg ): Low dose ketamine (sub-anesthetic) 0.5 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Ketamine (0.5 mg/kg): (sub-anesthetic) 0.5 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
- Ketamine (1 mg/kg): High dose (sub-anesthetic) 1 mg/kg ketamine following induction of anesthesia or administration of sedative medications.
  Ketamine (1 mg/kg): High dose (sub-anesthetic) 1 mg/kg ketamine following induction anesthesia or administration of sedative medications.
Arm/Group | Ketamine (0.5 mg/kg ) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Number analyzed (Participants) | 227 | 222 | 223
participants
  VAS day 1 | 70 [40 to 87] | 63.5 [43 to 82] | 68 [37.5 to 90]
  VAS day 2 | 56 [30 to 80] | 59 [31 to 80] | 57.5 [27 to 81]
  VAS day 3 | 46 [22.5 to 75] | 52.5 [25.5 to 75] | 47 [23 to 74]
  BPS/BPS-NI day 1 | 4 [3 to 5] | 4 [3 to 4] | 4 [3 to 5]
  BPS/BPS-NI 2 | 4 [3 to 4] | 3 [3 to 4] | 3 [3 to 4]
  BPS/BPS-NI 3 | 3 [3 to 4] | 3 [3 to 4] | 3 [3 to 4]
Statistical Analysis 1: Comparison: Ketamine (0.5 mg/kg ) vs Normal Saline (Placebo); We compared the combined average pain level (pain level at rest, taking a deep breath, and/or when moving) over the entire day (AM and PM); Test type: Superiority; p = 0.964, ANOVA; one-way

3. Secondary Outcome: Median Opioid Consumption
Description: Assessed from patients' medical charts. All morphine equivalent drugs consumed by patients perioperatively
  Opioid Drugs included:
  * Postoperatively while still in hospital, the list of pain medication used included Morphine, Hydromorphone, Meperidine, Nalbuphine, Oxycodone,Oxymorphone, Tramadol, bupivacaine, (Codeine, Fentanyl, Naloxone) Total Opiates (Morphine Equivalent) in milligrams The median(IQR) opioid consumption was compared across the three study groups Placebo vs. Lo-K (0.5 mg/kg) vs. Hi-K (1 mg/kg)
Time Frame: Postoperative days 0-3
Measure: Median (Full Range); unit: mg
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Number analyzed (Participants) | 227 | 222 | 223
mg | 88.9 [46.5 to 175.5] | 94.7 [48 to 199] | 78.7 [43.8 to 169]
Statistical Analysis 1: Comparison: Ketamine (0.5 mg/kg) vs Normal Saline (Placebo) vs Ketamine (1 mg/kg); All morphine equivalent drugs consumed by patients perioperatively Opioid Drugs included: * Postoperatively while still in hospital, the list of pain medication used included Morphine, Hydromorphone, Meperidine, Nalbuphine, Oxycodone,Oxymorphone, Tramadol, bupivacaine, (Codeine, Fentanyl, Naloxone) Total Opiates (Morphine Equivalent) in milligrams The median(IQR) opioid consumption was compared across the three study groups Placebo vs. Lo-K (0.5 mg/kg) vs. Hi-K (1 mg/kg); Test type: Superiority; p = 0.476, ANOVA

4. Secondary Outcome: Number of Patients With Postoperative Nausea and Vomiting
Description: Assessed from patient-reported postoperative nausea and vomiting section of Behavioral Pain Scale or Behavioral Pain Scale (Non-Intubated) Patients where asked whether they "currently have nausea/vomiting" AM & PM the response choices: None, Mild, Moderate, Severe Incidence of nausea\vomiting accounted for any positive reporting(Mild, moderate, or sever) Daily incidence accounted for any positive incidence AM/PM in each POD Any POD nausea/vomiting reports the incidence across day 1-3
  The incidence of nausea and or vomiting was compared across the three study groups Placebo vs. Lo-K (0.5 mg/kg) vs. Hi-K (1 mg/kg) for POD 1-3 and overall.
Time Frame: Postoperative days 1-3
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Number analyzed (Participants) | 227 | 222 | 223
Participants | 72 | 73 | 64
Statistical Analysis 1: Comparison: Ketamine (0.5 mg/kg) vs Normal Saline (Placebo); Assessed from patient-reported postoperative nausea and vomiting section of Behavioral Pain Scale or Behavioral Pain Scale (Non-Intubated) Patients where asked whether they "currently have nausea/vomiting" AM & PM the response choices: None, Mild, Moderate, Severe Incidence of nausea\vomiting accounted for any positive reporting(Mild, moderate, or sever) Daily incidence accounted for any positive incidence AM/PM in each POD Any POD nausea/vomiting reports the incidence across day 1-3; Test type: Superiority; p = 0.572, Chi-squared; frequency-test = 0.572

5. Secondary Outcome: ICU and/or Hospital Length of Stay
Description: Assessed from patients' medical charts
Time Frame: Postoperative period
Population: Outcome measure data were not collected.
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Adverse Outcomes (Number of Patients With Hallucinations)
Description: Assessed via Confusion Assessment Method or Confusion Assessment Method for Intensive Care Unit
Time Frame: Postoperative days 1-3
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Number analyzed (Participants) | 227 | 222 | 223
Participants | 45 | 40 | 62
Statistical Analysis 1: Comparison: Ketamine (0.5 mg/kg) vs Normal Saline (Placebo) vs Ketamine (1 mg/kg); Frequency of patients reporting hallucinations using the DSAQ instrument; Test type: Superiority; p = 0.01, Chi-squared

7. Secondary Outcome: Adverse Outcomes (Number of Patients With Nightmares)
Description: Assessed via Confusion Assessment Method or Confusion Assessment Method for Intensive care Unit
Time Frame: Postoperative days 1-3
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
Number analyzed (Participants) | 227 | 222 | 223
Participants | 27 | 18 | 34
Statistical Analysis 1: Comparison: Ketamine (0.5 mg/kg) vs Normal Saline (Placebo) vs Ketamine (1 mg/kg); Test type: Superiority; p = 0.03, Chi-squared — Patients where asked whether "Following their surgery they had bad dreams or nightmares the response choices: Yes/No question The incidence of hallucination and nightmares were assessed separately and compared across the three study group

ADVERSE EVENTS:
Time Frame: Assessed up to 3 days (POD 0-3).
Arm/Group | Ketamine (0.5 mg/kg) | Normal Saline (Placebo) | Ketamine (1 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/227 | 2/220 | 0/223
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/222 | 0/223
Other Adverse Events (participants affected / at risk) | 90/227 | 82/222 | 86/223
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (0.5 mg/kg) (N=227) | Normal Saline (Placebo) (N=222) | Ketamine (1 mg/kg) (N=223)
Atrial Fibriliation (Nervous system disorders) | 21 (21) | 19 (19) | 15 (15)
Anaemia/Bleeding (Blood and lymphatic system disorders) | 19 (19) | 13 (13) | 20 (20)
Infection (Infections and infestations) | 16 (16) | 18 (18) | 15 (15)
Renal (Renal and urinary disorders) | 13 (13) | 11 (11) | 8 (8)
Hypotension (Vascular disorders) | 11 (11) | 11 (11) | 9 (9)
Tachycardia (Cardiac disorders) | 8 (8) | 8 (8) | 8 (8)
Gastrointestinal (Gastrointestinal disorders) | 9 (9) | 8 (8) | 6 (6)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No